CLINICAL TRIAL: NCT00758251
Title: Observation of Change in Clinical Global Impression Scores in Schizophrenia Patients Receiving Seroquel XR Treatment
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Janis Dobelis, Country Manager, AstraZeneca MC Latvia
Other Study IDs: NIS-NLV-SER-2008/1
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Seroquel XR; CGI
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Adult schizophrenia patients already on Seroquel XR therapy

SUMMARY:
The purpose of this study is to assess severity of illness in schizophrenia patients in routine clinical practice at the time of entry in the study and after the treatment with Seroquel XR for 8 weeks.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Schizophrenia prescribed on Seroquel XR according to the approved product information before inclusion in this non-interventional study
* Signed and dated Patient Informed Consent (ICF)

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients of Seroquel XR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Improvement in CGI scores and BPRS comparing visits 1 and 3. | twice with 4 week interval

SECONDARY OUTCOMES:
To evaluate compliance to therapy | twice with 4 week interval

CONTACTS AND LOCATIONS:
Overall Officials: Agrita Hartmane, Study Director — AstraZeneca Latvia
Locations (15):
- Latvia (15):
  - Research Site, Bauska
  - Research SIte, Cēsis
  - Research Site, Daugavpils
  - Research Site, Dobele
  - Research Site, Jelgava
  - Research Site, Jēkabpils
  - Research Site, Jūrmala
  - Research Site, Kuldīga
  - Research Site, Liepāja
  - Research Site, Riga
  - Research Site, Saldus
  - Research Site, Strenči
  - Research Site, Talsi
  - Research Site, Tukums
  - Research Site, Valmiera